## **Informed Consent forms**

# Official title: Novel Therapies in Moderately Severe Acute Alcoholic Hepatitis

NCT number: NCT01922895

IRB Approved date: September 13, 2017

## The University of Texas Southwestern Medical Center at Dallas Parkland Health & Hospital System

#### **CONSENT TO PARTICIPATE IN RESEARCH**

Title of Research: Novel therapies in moderately severe alcoholic hepatitis

Funding Agency/Sponsor: NIH (funded)

Study Doctors: Mack Mitchell, M.D.

Lisa Casey, M.D. Jennifer Cuthbert, M.D.

Study Personnel

Co-Investigator: Blair Holbein, Ph.D.

You may call these study doctors or research personnel during regular office hours at 214-648-4570. At other times, you may call them at 214-648-3111 and tell them that you need to contact your study doctors. Have the study information with you when you call after hours so that the hospital operators know who to contact.

#### Instructions:

Please read this consent form carefully and take your time making a decision about whether to participate. As the researchers discuss this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. The purpose of the study, risks, inconveniences, discomforts, and other important information about the study are listed below. If you decide to participate, you will be given a copy of this form to keep.

#### What you should know about this study:

- You are being asked to join a research study.
- This consent form explains the research study and your part in the study.
- Please read it carefully and take as much time as you need.
- Please ask questions at any time about anything you do not understand
- You are a volunteer. If you join the study, you can change your mind later. You can
  decide not to take part or you can quit at any time. There will be no penalty or loss of
  benefits if you decide to quit the study.
- If you are not scheduled to undergo a procedure for clinical reasons, you must be an adult with the capacity to give consent in order to provide blood or spinal fluid.
- During the study we will tell you if we learn any new information that might affect whether you wish to continue to be in the study.
- Ask your study doctor or the study team to explain any words or information in this informed consent that you do not understand.





#### Why is this research being done?

The purpose of this study is to start an electronic database for patient information and to collect blood, tissue and other samples from people, being evaluated or treated for liver inflammation (hepatitis) from alcohol.

We are collecting these samples and medical information so that they can be made available to research scientists who are involved in the study of these diseases. This research is attempting to improve upon our ability to diagnose these conditions.

#### What will happen if you join this study?

If you agree to be in this study, we will ask you to do the following things:

<u>Medical Record Review</u>: Your medical records will be reviewed by a member of our team and selective data will be entered into a secure electronic database. This will include history and physical examination, results of x-rays, pathology, blood counts, clotting, and chemistry tests for the liver. Medical records will be reviewed on a regular basis to ensure up to date information.

<u>Specimen Samples</u>: If as part of your clinical care, a blood draw or biopsy is performed, some of the fluid or tissue will be placed into our repository for future research studies. You may also be asked to consent to a blood draw to collect samples solely for research purposes (only if you are an adult with capacity to give consent). You do not need to provide these samples to be part of the database.

For identification purposes, you will be assigned a coded identifier and will not be personally identifiable. This code will be placed on all the material that is sent to the research laboratories.

Information about your medical history, portions of samples and results of tests may be shared with national and international research partners and may be entered into secondary national and international databases. The sharing of this information is meant to increase collaborative projects and bolster worldwide research efforts. The information provided to them will not include your name, medical record number or unique identifiers. It may include your age, date of birth, city of residence or dates of tests.

#### Will I be contacted again?

Yes, you may also be contacted if updated medical information is needed for the database.

#### Will my specimen be stored for future use?

Yes, your blood specimens or other samples will be evaluated by research scientists studying various liver diseases. Some portion may be frozen or stored indefinitely for this future use. Stored specimens may be analyzed in the future using additional technologies without you being asked to sign another consent form.

## Will my samples be used to study any other diseases besides my condition?

Yes. An important part of this research is to allow for associations to be made between different diseases. Your sample may be used for broad-based research for a variety of disease states.

## Will my sample be used for genetic research?






Study ID: STU 092012-012 Date Approved: 9/13/2017

Yes. Genetic research is an important part of the investigation into the causes of these diseases. The causes of many of these diseases are believed to be the result of combinations of inherited genes and possible various exposures to the environment. Genetic research is an important part of the investigation into the causes of these diseases. There are no plans to inform you, or your relatives, about the results of genetic studies, since at this time the information is not thought to be medically useful.

#### What is DNA?

DNA means *deoxyribonucleic acid*. DNA is the substance in our cells which contains information we inherited from our parents and other family members. Your DNA contains "genes" which predict things like physical characteristics (eye color, hair color, height, etc.) and may also be a factor in whether you develop or are at risk of developing certain illnesses or disorders.

**How is DNA obtained?** Cells from blood or other body materials are processed in a laboratory that has special equipment that can extract DNA and identify genes.

## What are the risks or discomforts of the study?

There is a risk that your personal health information could be seen by people not working on the study.

The risks of a blood draw include pain, bruising and same patients have lost consciousness during the process.

Collection of the Tissue Samples: You may undergo a liver biopsy for your liver disease. If this is planned, your doctor will have discussed this with you. This procedure has been deemed medically necessary and you have agreed to the procedure. Participation in this research will mostly involve using what is called "medical waste." Medical waste is leftover tissue that is not needed for diagnosis of your liver disease.

Because all specimens obtained for research will come from your routinely scheduled procedures, there will be no additional risk or discomfort related to participating in this research. The only potential risk to you is accidental release of your medical information.

## Problems obtaining insurance or employment

A new Federal Law called the Genetic Information Nondiscrimination Act of 2008 (GINA), generally makes it illegal for group and individual health insurers from using your genetic information to set insurance eligibility, premiums, or contribution amounts. They cannot request or require that you take a genetic test. In addition, employers with 15 or more employees may not use your genetic information to make decisions regarding hiring, firing, job assignments, or promotions, nor can they request, require, or purchase your genetic information. GINA does not protect you against genetic discrimination by companies that sell life, disability, or long-term care insurance.

#### Are there risks related to pregnancy?

The risks in pregnancy are the same as the general risks of the study, outlined above. Patients who are concerned about their pregnancy should discuss any concerns with their obstetrician before taking part in the study.


DO NOT FILE OR SCAN THIS CONSENT FORM INTO THE MEDICAL RECORD



## What should I do if I think I am having problems?

If you have unusual symptoms, pain, or any other problems while you are in the study, you should report them to the researchers right away. Telephone numbers where they can be reached are listed on the first page of this consent form.

If you have a sudden, serious problem, like difficulty breathing or severe pain, go to the nearest hospital emergency room, or call 911 (or the correct emergency telephone number in your area). Tell emergency personnel about any medications you are taking, including any medications you are taking for this study.

#### Are there benefits to being in the study?

There will be no direct medical benefit to you. Since it is possible that the causes of one, some or all of the liver diseases could be determined because of research using your samples, someone may benefit in the future.

## What are your options if you do not want to be in the study?

You do not have to join this study. If you do not join, your care will not be affected.

## Will it cost you anything to be in this study?

No.

## Will you be paid if you join this study?

No.

## Can you leave the study early?

Yes. You may withdraw your consent by contacting your study doctor, Dr. Mitchell at 214-648-4570 during regular business hours and at 214-648-3111 after hours and on weekends and holidays. However, samples that have been already used for research, as well as any results or information already collected before you withdraw from the study, cannot be destroyed. Refusing to take part in the future will not affect your current or future medical care in any way. If you withdraw from this study at any time, we will stop contacting you.

## Will my information be kept confidential?

Medical information collected during this study and the results of any test or procedure done may be included in your medical record and this information may be available to health care providers and authorized persons including your insurance company.

You should know that certain organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- Cleveland Clinic, University of Louisville, University of Massachusetts, NIH
- Representatives of government agencies, like the U.S. Food and Drug Administration (FDA), involved in keeping research safe for people; and
- The UT Southwestern Institutional Review Board.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.




In addition to this consent form, you will be asked to sign an "Authorization for Use and Disclosure of Protected Health Information." This authorization will give more details about how your information will be used for this research study, and who may see and/or get copies of your information.

If you do cancel your permission to use and disclose your information, your part in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in this study.

## What will happen if I am harmed as a result of taking part in this study?

Compensation for an injury resulting from your participation in this research is not available from the University of Texas Southwestern Medical Center at Dallas or Parkland Health & Hospital System.

You retain your legal rights during your participation in this research

What happens to Data, Tissue, Blood and Specimens that are collected in the study? Researchers at UT Southwestern work to find the causes and cures of disease. The data, tissue, blood and specimens collected from you during this study are important to both this study and to future research.

If you join this study:

- You will not own the data, or the tissue, blood, or other specimens given by you to the investigators for this research.
- Both UT Southwestern and any sponsor of this research may study your data and the tissue, blood, or other specimens collected from you.
- If data, tissue, blood, or other specimens are in a form that identifies you, UT Southwestern may use them for future research only with your consent or IRB approval.
- You will not own any product or idea created by the researchers working on this study.
- You will not receive any financial benefit from the creation, use or sale of such a product or idea.

RD



#### **SIGNATURES:**

#### YOU WILL BE GIVEN A COPY OF THIS CONSENT FORM TO KEEP.

Your signature below certifies the following:

- You have read (or been read) the information provided above.
- You have received answers to all of your questions and have been told who to call if you
  have any more questions.
- You have freely decided to participate in this research.
- You understand that you are not giving up any of your legal rights.
- You understand that a copy of this signed consent document, information about this study and the results of any test or procedure done may be included in your medical record and this information may be available to health care providers and authorized persons including your insurance company.

| Signature of Participant (18 yrs or older) | Printed Name of Participant (18 yrs or older) | Date | Time | AM/PM |
|---|---|---|---|---|
| NAME OF PERSON OBTAIN | IING CONSENT | | | |
| Signature | Printed Name | <br>Date | Time | AM/PM |



## The University of Texas Southwestern Medical Center at Dallas Parkland Health & Hospital System

#### CONSENT TO PARTICIPATE IN RESEARCH

Title of Research: Novel therapies in moderately severe alcoholic hepatitis

Funding Agency/Sponsor: NIH (funded)

Study Doctors: Mack Mitchell, M.D.

Lisa Casey, M.D.

Jennifer Cuthbert, M.D.

You may call these study doctors or research personnel during regular office hours at 214-648-4570. At other times, you may call them at 214-648-3111 and tell them that you need to contact your study doctors. Have the study information with you when you call after hours so that the hospital operators know who to contact.

#### Instructions:

Please read this consent form carefully and take your time making a decision about whether to participate. As the researchers discuss this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. The purpose of the study, risks, inconveniences, discomforts, and other important information about the study are listed below. If you decide to participate, you will be given a copy of this form to keep.

#### Why is this study being done?

This study is being done to find out whether supplementing your diet, with a special nutrient, can treat your condition better or more safely than standard medicine.

#### Why is this considered research?

This is a research study because the dietary supplement is not recognized for the treatment of patients with liver problems.

## The following definitions may help you understand this study:

- Double-blind means neither you nor the researchers will know which drug you are receiving.
- Placebo-controlled means that some participants will get a placebo. A placebo looks like the investigational drug but it includes no active ingredients.
- Randomization means you will be placed by chance (like a flip of a coin) in one of the study groups.
- Standard medical care means the regular care you would receive from your personal doctor if you choose not to participate in this research.



 Researcher means the study doctors and research personnel at the University of Texas Southwestern Medical Center at Dallas and its affiliated hospitals.

## Why am I being asked to take part in this research study?

You are being asked to take part in this study because you have an inflamed liver (hepatitis) that your doctors' think is from your body's reaction to alcohol.

## Do I have to take part in this research study?"

No. You have the right to choose whether you want to take part in this research study. If you decide to participate and later change your mind, you are free to stop participation at any time. If you decide not to take part in this research study it will not change your legal rights or the quality of health care that you receive at this center.

## How many people will take part in this study?

About 50 people will take part in this study at UT Southwestern or Parkland Health and Hospital System. This study also is taking place at a number of other medical facilities around the country. There will be a total of 130 people participating in this research study throughout the United States.

## What is involved in the study?

If you volunteer to take part in this research study, you will be asked to sign this consent form and will have the following tests and procedures. Some of the procedures may be part of your standard medical care, but others are being done solely for the purpose of this study.

## Screening Procedures

To help decide if you qualify to be in this study, the researchers will ask you questions about your health, including medications you take, your diet and habits. They will also get information from your medical record.

### **Group Assignment**

If the researchers believe you can take part in this study, you will be assigned randomly (like a flip of a coin) to receive either an active diet supplement or an inactive one (a placebo).

For 6 months, everyone gets an identical-appearing supplement. If the researchers knew which patients were getting the study drug they might be tempted to favor it.

All study supplements will finish after 6 months.

The group you will be in is decided by your study number. This is linked to instructions that are kept in the hospital pharmacy. The pharmacy will provide you with your medications when you are in the hospital and also give you your medications to take at home. Neither you nor the researchers will be allowed to choose which group you are assigned to; neither you nor the researchers will know which group you are in.



## Study Medication/Intervention

If you decide to participate in this study you will take a supplement to your diet every day for 6 months. The supplement is Culturelle (Lactobacillus Rhamnosus GG).

## <u>Procedures and Evaluations during the Research</u>

All study subjects will receive the standard medical care used for hepatitis from your body's reaction to alcohol. This includes:

- 1. A good diet while in the hospital and recommendations for what to eat at home
  - a. Lots of fresh vegetables, fruits, chicken, fish
  - b. Vitamins and other special nutrition if needed
- 2. Help with avoiding alcohol in the future
  - a. Counselors
  - b. Psychologists
  - c. Rehabilitation assistance
- Only take medications prescribed by your doctors. Do not take any medication or diet supplement or over-the-counter remedy without checking with a study doctor or nurse. Avoid all pain medicines that have high risk associated with them because of liver disease.
  - a. Aspirin and over the counter medications like ibuprofen Motrin®, Aleve® can damage the kidneys with as little as one tablet
  - b. Stronger pain medicines that contain codeine or a similar agent can cause confusion related to liver disease
  - c. Acetaminophen (Tylenol®) can directly cause liver damage
- 4. Treatment for any complications that can occur
  - a. Antibiotics for infections
  - b. Treatment for diarrhea or constipation or nausea and vomiting if they occur
- 5. Blood drawing to follow the changes in your liver.
- 6. Follow-up in the regular outpatient liver clinic, after you leave the hospital, until your liver has completely recovered. The number of visits depends on how quickly you get better. This is likely to be:
  - a. 1 week after leaving the hospital
  - b. 1-2 visits in the next month
  - c. 1-2 visits in the next 2-4 months, depending on how quickly you get well
  - d. A final clinic visit after 6 months

In addition, the following special, extra studies will be done for research purposes:

| Where | When | | What | How |
|---|---|---|---|---|
| In hospital | First of study | day | Inflammation markers and liver | Research tests: Taking extra tubes of blood |
| | | | condition. A nutritional assessment with a hand grip dynamometer. | blood tests (amount = 3 |



| | | Blood, stool, and urine for testing to see why alcohol caused your body to react in this way. These tests are done as part of the standard treatment for your condition. | |
|---|---|---|---|
| In clinic | 7 day<br>1 month<br>3 months<br>6 months | Inflammation markers and liver markers will be measured. These tests are done as part of the research on treatment for your condition. Blood and urine for testing to see why alcohol caused your body to react in this way. These tests are done as part of the standard treatment for your condition. | Taking extra tubes of blood when you have regular blood tests (amount = 3 tablespoons). Collecting urine and stool in a container. |

The inflammation and liver markers in this study are designed for research, not for medical purposes. They are not useful for finding problems or diseases. Even though the researchers are not looking at your inflammation and liver markers to find or treat a medical problem, you will be told if they notice something unusual. You and your regular doctor can decide together whether to follow up with more tests or treatment. Because the inflammation and liver markers done in this study are not for medical purposes, the research results will not be sent to you or to your regular doctor. Your anonymous sample will be sent to coordinating research centers outside of UT Southwestern who are studying your disease. Your sample will be made anonymous by removing any identifiable information about you before it is shared with investigators outside of UT Southwestern.

#### Study Procedures by Study Day:

A summary of evaluations is located in the schedule of events table provided at the end of this section. The procedures and evaluations are outlined below.

#### Screening:

Complete screening will occur once the informed consent has been obtained as described above. Individuals who are not eligible for the study will be given the option for the same follow-up without the study medicine.

The study subject's general health and study information include:

- Signed consent
- Other routine information including sex, date of birth, race and ethnic group (Hispanic or not).



- Medicine history over the past 30 days, including prescribed and over-the-counter ones, herbal remedies, vitamins and minerals.
- Alcohol in the past 60 days and for the years before.
- Drawing blood for blood counts, clotting, and chemistry tests for the liver, pancreas and kidneys; female study subjects will have a pregnancy test. These are standard tests for your condition. The total amount of blood for these tests is about 7 tablespoons.
- Physical examination, including height, weight, and vital signs (blood pressure, pulse, breathing and temperature)
- Imaging of the abdomen.

## Assessments at baseline and during study treatment:

Study Procedures by Study Day:

A summary is in the table at the end of this section.

Study day 0 – start (within 48 hours of study beginning)

- · Record health history and review alcohol use.
- Standard of care laboratory studies (chemistry, blood count, clotting, urine, infection including tuberculosis testing).
- Tests for fluid in belly, if it is there
- Nutritional Assessment with a hand grip measurement.
- Urine, blood (3 tablespoons) and stool testing for research.
- Make a list of all medicines including those purchased over the counter, from health food stores and other remedies.
- Check blood pressure, pulse, temperature and breathing (vital signs) and physical exam.

## Treatment day 1 – time zero

- Begin study medicine once daily.
- Standard blood tests for your condition (1 tablespoon)

## Treatment day 2:

- Inpatient assessment to include:
  - Review health history for changes.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine and ½ tablespoon of blood).
  - 24 hour urine collection.
- Continue study medicine once daily.
- Standard blood tests for your condition (1½ tablespoons)

## Treatment days 3-6:

If study subject remains inpatient or has outpatient visit:



- Review health history for changes. .
- List all medicines
- Check vital signs and physical exam
- Continue study medicine once daily.
- Standard blood tests for your condition (1 tablespoon)

## Treatment day 7 ± 2 days:

- Inpatient assessment or **required** outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine and 2 tablespoon of blood).
- · Continue study medicine once daily.
- Standard and research blood tests (2 tablespoons)
  - Nutritional Assessment with hand grip measurement.

## Treatment days 8-14:

- If study subject remains inpatient or has outpatient visit:
  - Review health history for changes. Review alcohol intake.
  - · List all medicines
  - Check vital signs and physical exam
- Continue study medicine once daily.
- Standard blood tests for your condition (1 tablespoon)

#### Treatment days 15-27:

- If study subject remains inpatient or has a clinically indicated outpatient visit:
  - Review health history for changes. Review alcohol intake.
  - · List all medicines
  - Check vital signs and physical exam
- · Continue study medicine once daily.
- Standard blood tests for your condition (1 tablespoons)

## Treatment day 28 ± 2 days:

- Inpatient assessment or **required** outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine and 3 tablespoon blood).
- · Continue study medicine once daily.
- Standard and blood tests for your condition (1½ tablespoon)
  - Nutritional Assessment with hand grip measurement

## Treatment day 29 to 2 months:

Continue study medicine once daily.



- If study subject remains inpatient during this interval or completes clinically indicated outpatient visit during this time, the following data will be recorded:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Standard blood tests for your condition (1 tablespoons)

## Treatment 3 months ± 2 weeks:

- Inpatient assessment or required outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine, stool, and 3 tablespoon blood).
- Continue study medicine once daily
- Standard blood tests for your condition (1½ tablespoon)

#### Treatment 4, 5 months ± 2 weeks:

- Continue study medicine once daily
- If study subject remains inpatient or completes clinically indicated outpatient visit during this time, the following will be done:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - · Check vital signs and physical exam
  - Standard blood tests for your condition (1 tablespoons)

#### Treatment 6 months ± 2 weeks:

- STOP study medicines.
- Complete abdominal ultrasound.
- Inpatient assessment or **required** outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine, 3 tablespoon blood and stool).
- Standard blood tests for your condition (1½ tablespoons)
  - Nutritional Assessment with hand grip measurement

## Follow up of early end of study:

A safety visit will be done about 30 days after stopping of study medicine for all study subjects who stopped before the end. This will include:

- Standard blood tests for your condition (chemistry, blood count and clotting).
- Check vital signs and physical exam
- Review health history for changes. Review alcohol intake.
- List all medicines
- Review reason for early stopping.
- Standard and research blood tests (2 tablespoons total)



| Purpose | Test | Day 0 | Day 2 – 6* | Day 7 | Day<br>8 – 27* | Day<br>28 | 2 mos* | 3 mos | 4 mos* | 5 mos* | 6 mos |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Standard | General health and liver questions | х | х | х | х | х | х | х | х | х | х |
| | Questions about drinking alcohol | х | х | х | х | х | х | х | х | х | х |
| | Physical exam | х | х | х | х | х | х | х | х | х | х |
| Blood | Liver tests | х | х | х | х | х | х | х | х | х | х |
| | Tests of chemicals and kidneys | х | х | х | х | х | х | х | х | х | Х |
| | Blood count | х | х | х | х | х | х | х | х | х | Х |
| | Cholesterol test | х | | | | | | | | | х |
| | Pancreas tests | х | | | | | | | | | |
| | Tests for viruses and bacteria | х | | | | | | | | | |
| | TB skin test | х | | | | | | | | | |
| Urine | Urine tests | х | | | | | | | | | |
| | Poisons | х | | | | | | | | | |
| Fluid | Belly fluid chemicals and infection | х | | | | | | | | | |
| Stool | Infection tests | х | | | | | | | | | |
| Imaging | Ultrasound of belly | х | | | | | | | | | х |
| Research | Gut leakiness | х | | | | х | | х | | | х |
| | Zinc levels | х | | | | х | | х | | | х |
| | Stool bacteria tests | х | | | | | | х | | | х |
| | Inflammation tests | х | x-day 2 | х | | х | | х | | | х |

<sup>\*</sup> if clinically indicated



## <u>Procedures for storing of extra or left over samples</u>

Samples of your blood and urine will be frozen and stored so that the researchers can test for any new inflammation or liver markers that are developed.

- Samples will be labeled with a study number, not with your name or other personal number.
- The key for study numbers will be kept in your medical record in a special section for research study information.
- The anonymous samples will be sent to Cleveland Clinic for storage
- The Principal Investigators will decide where and how the remaining samples will be processed
- Samples may be sent to other scientists for studies approved by their local IRB's to further understand this disease.

## How long can I expect to be in this study?

The study is for a total of 6 months, 6 months on tablets. You can choose to stop participating for any reason at any time. However, if you decide to stop participating in the study, we encourage you to tell the researchers. You will be asked if you are willing to complete some study termination tests.

## What are the risks of the study?

Study Procedure/Intervention

Because of your participation in this study, you are at risk for the following side effects. You should discuss these with the researchers and your regular health care provider.

**Dietary Supplement (Probiotics):** Bacteria are normally found in the gastrointestinal tract. They are deliberately cultured in yogurts and are a nutritional supplement.

| Side effects | Frequent | Occasional | Rare |
|---|---|---|---|
| Side effects | >20% of subjects | 2 - 20% of subjects | Less than 2% of subjects |
| Serious | | | Infection with probiotic |
| | | | bacteria (1 adult) |
| Less Serious | | | |
| Minor | | Burping | |
| | | Hiccups | |

## Psychological Stress

Some of the questions we will ask you about your personal habits, as part of this study, may make you feel uncomfortable. You may refuse to answer any of the questions, take a break or stop your participation in this study at any time.

## Loss of Confidentiality

Any time information is collected; there is a potential risk for loss of confidentiality.



Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

## Risks of Blood Drawing

Risks associated with drawing blood from your arm include minimal discomfort and/or bruising. Infection, excess bleeding, clotting, and/or fainting also are possible, although unlikely. You will have You will have 6 tablespoons of blood collected because you are in this research study, in addition to the tests that you need to take care of your health (another 13 tbspns over the 6 months).

## Other Risks

There may possibly be other side effects that are unknown at this time. If you are concerned about other, unknown side effects, please discuss this with the researchers.

## How will risks be minimized or prevented?

Potential risks and discomforts will be minimized to the greatest extent possible by appropriate training of all researchers and study personnel, monitoring you closely, withdrawal from the study upon evidence of difficulty or an adverse event; referral for treatment, counseling or other necessary follow-up.

## What will my responsibilities be during the study?

While you are part of this study, the researchers will follow you closely to determine whether there are problems that need medical care. It is your responsibility to do the following:

- Ask questions about anything you do not understand.
- Keep your appointments.
- Follow the researchers' instructions.
- Let the researchers know if your telephone number or address changes.
- Store study tablets in a secure place at home away from anyone who is unable to read and understand labels, especially children.
- Tell the researchers before you take any new medication, even if it is prescribed by another doctor for a different medical problem or something purchased over the counter.
- Tell your regular doctor about your participation in this study.
- Carry information about contacting the study doctors in your purse or wallet.
- Report to the researchers any injury or illnesses while you are on study, even if you do not think they are related.

## If I agree to take part in this research study, will I be told of any new risks that may be found during the course of the study?

Yes. You will be told if any new information becomes available during the study that could cause you to change your mind about continuing to participate or that is important to your health or safety.

Study ID: STU 092012-012 Date Approved: 9/13/2017



## What should I do if I think I am having problems?

If you have unusual symptoms, pain, or any other problems while you are in the study, you should report them to the researchers right away. Telephone numbers where they can be reached are listed on the first page of this consent form. If you have a sudden, serious problem, like difficulty breathing or severe pain, go to the nearest hospital emergency room, or call 911 (or the correct emergency telephone number in your area). Tell emergency personnel about any medications you are taking, including any medications you are taking for this study.

## What are the possible benefits of this study?

If you agree to take part in this study, there may or may not be direct benefits to you. The researchers cannot guarantee that you will benefit from participation in this research. We hope that the information learned from this study will benefit others with inflammation of the liver from alcohol. Information gained from this research could lead to treatment with lower risks of dying in the first 6 months after being admitted to the hospital for hepatitis from alcohol.

## What options are available if I decide not to take part in this research study?

You do not have to participate in this research to receive care for your medical problem. Instead of being in this study, you have the following option:

 Standard of care treatment through abstinence from alcohol and general supportive care (nutritional support and hydration)

Please talk to the researchers or your personal doctor about these options.

## Will I be paid if I take part in this research study?

There are no funds available to pay for parking expenses, transportation to and from the research center, lost time away from work etc., lost wages, or child care expenses.

## Will my insurance provider or I be charged for the costs of any part of this research study?

No. Neither you, nor your insurance provider, will be charged for anything done only for this research study. However, the standard medical care for your condition (care you would have received whether or not you were in this study) is your responsibility (or the responsibility of your insurance provider or governmental program). You will be charged, in the standard manner, for any procedures performed for your standard medical care.

## What will happen if I am harmed as a result of taking part in this study?

It is important that you report any illness or injury to the research team listed at the top of this form immediately. Compensation for an injury resulting from your participation in this research is not available from the University of Texas Southwestern Medical Center or Parkland Health & Hospital System. You retain your legal rights during your participation in this research



## Can I stop taking part in this research study?

Yes. If you decide to participate and later change your mind, you are free to stop taking part in the research study at any time. If you decide to stop taking part in this research study, it will not affect your relationship with the UT Southwestern staff or doctors. Whether you participate or not will have no effect on your legal rights or the quality of your health care.

## If I agree to take part in this research study, can I be removed from the study without my consent?

Yes. The researchers may decide to take you off this study if:

- Your medical problem becomes worse.
- The researchers believe that participation in the research is no longer safe for vou.
- You are unable to follow the researcher's instructions.

## Will my information be kept confidential?

Medical information collected during this study and the results of any test or procedure done may be included in your medical record and this information may be available to health care providers and authorized persons including your insurance company.

You should know that certain organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- · Cleveland Clinic, University of Louisville, University of Massachusetts, NIH
- Representatives of government agencies, like the U.S. Food and Drug Administration (FDA), involved in keeping research safe for people; and
- The UT Southwestern Institutional Review Board.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by the U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

In addition to this consent form, you will be asked to sign an "Authorization for Use and Disclosure of Protected Health Information." This authorization will give more details about how your information will be used for this research study, and who may see and/or get copies of your information.

Are there procedures I should follow after stopping participation in this research? Yes. If you, the researchers, or the sponsor stops your participation in the research, you may be asked to do the following:

 Let the researchers know immediately that you wish to withdraw from the research.



- Return to the research center for tests that may be needed for your safety.
- Return any unused study materials, including empty containers.
- Discuss your future medical care, if any, with the researchers and/or your personal doctor.

#### Whom do I call if I have questions or problems?

For questions about the study, contact Dr. Mitchell at 214-648-4570 during regular business hours and at 214-648-3111 after hours and on weekends and holidays.

For questions about your rights as a research participant, contact the UT Southwestern Institutional Review Board (IRB) Office at 214-648-3060.

#### **SIGNATURES:**

#### YOU WILL BE GIVEN A COPY OF THIS CONSENT FORM TO KEEP.

Your signature below certifies the following:

- You have read (or been read) the information provided above.
- You have received answers to all of your questions and have been told who to call if you have any more questions.
- You have freely decided to participate in this research.
- You understand that you are not giving up any of your legal rights.
- You understand that a copy of this signed consent document, information about this study and the results of any test or procedure done may be included in your medical record and this information may be available to health care providers and authorized persons including your insurance company.

| Participant's Name (printed) | |
|------------------------------|-------------|
| Tantopanto Namo (printoa) | |
| Participant's Signature | Date & Time |



| Name of person obtaining consent (printed) | |
|--------------------------------------------|-------------|
| Signature of person obtaining consent | Date & Time |

MEDICAL COUNTY

## The University of Texas Southwestern Medical Center at Dallas Parkland Health & Hospital System

#### **CONSENT TO PARTICIPATE IN RESEARCH**

Title of Research: Novel therapies in moderately severe alcoholic hepatitis

Funding Agency/Sponsor: NIH (funded)

Study Doctors: Mack Mitchell, M.D.

Lisa Casey, M.D.

Jennifer Cuthbert, M.D.

You may call these study doctors or research personnel during regular office hours at 214-648-4570. At other times, you may call them at 214-648-3111 and tell them that you need to contact your study doctors. Have the study information with you when you call after hours so that the hospital operators know who to contact.

#### Instructions:


Please read this consent form carefully and take your time making a decision about whether to participate. As the researchers discuss this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. The purpose of the study, risks, inconveniences, discomforts, and other important information about the study are listed below. If you decide to participate, you will be given a copy of this form to keep.

## Why is this study being done?

This study is being done to follow what happens to the liver in response to inflammation from alcohol by collecting and testing research samples. The research studies will not improve the health of your liver.

## Why is this considered research?

This is a research study because the tests are not routine for patients with liver problems.

### The following definitions may help you understand this study:

- Standard medical care means the regular care you would receive from your personal doctor if you choose not to participate in this research.
- Researcher means the study doctors and research personnel at the University of Texas Southwestern Medical Center at Dallas and its affiliated hospitals.

## Why am I being asked to take part in this research study?

You are being asked to take part in this study because you have an inflamed liver (hepatitis) that your doctors' think is from your body's reaction to alcohol.

Do I have to take part in this research study?

DO NOT DISCLOSE





Study ID: STU 092012-012 Date Approved: 9/13/2017

No. You have the right to choose whether you want to take part in this research study. If you decide to participate and later change your mind, you are free to stop participation at any time. If you decide not to take part in this research study it will not change your legal rights or the quality of health care that you receive at this center.

#### How many people will take part in this study?

About 50 people will take part in the medication study at UT Southwestern or Parkland Health and Hospital System. This study also is taking place at a number of other medical facilities around the country. There will be a total of 130 people participating in this research study throughout the United States. People who don't want to take a medication can be part of the research by participating in the new tests.

## What is involved in the study?

If you volunteer to take part in this research study, you will be asked to sign this consent form and will have the following tests and procedures. Some of the procedures may be part of your standard medical care, but others are being done solely for the purpose of this study.

## Screening Procedures

To help decide if you qualify to be in this study, the researchers will ask you questions about your health, including medications you take, your diet and habits. They will also get information from your medical record.

## Procedures and Evaluations during the Research

All study subjects will receive the standard medical care used for patients with hepatitis from your body's reaction to alcohol. This includes:

- 1. A good diet while in the hospital and recommendations for what to eat at home
  - a. Lots of fresh vegetables, fruits, chicken, fish
  - b. Vitamins and other special nutrition if needed
- 2. Help with avoiding alcohol in the future
  - a. Counselors
  - b. Psychologists
  - c. Rehabilitation assistance
- 3. Only take medications prescribed by your doctors. Do not take any medication or diet supplement or over-the-counter remedy without checking with a study doctor or nurse. Avoid all pain medicines that have high risk associated with them because of liver disease.
  - a. Aspirin and over the counter medications like ibuprofen Motrin®, Aleve® can damage the kidneys with as little as one tablet
  - b. Stronger pain medicines that contain codeine or a similar agent can cause confusion related to liver disease
  - c. Acetaminophen (Tylenol®) can directly cause liver damage
- 4. Treatment for any complications that can occur
  - a. Antibiotics for infections
  - b. Treatment for diarrhea or constipation or nausea and vomiting if they occur
- 5. Blood drawing to follow the changes in your liver.
- 6. Follow-up in the regular outpatient liver clinic, after you leave the hospital, until your liver has completely recovered. The number of visits depends on how quickly you get better. This is likely to be:
  - a. 1 week after leaving the hospital

CONTINUES OF STREET OF STR

- b. 1-2 visits in the next month
- c. 1-2 visits in the next 2-4 months, depending on how quickly you get well
- d. A final clinic visit after 6 months

In addition, the following special, extra studies will be done for research purposes when you come into clinic:

| Where | When | | What | How |
|---|---|---|---|---|
| In<br>hospital | | day<br>the | Inflammation markers and liver markers will be measured. These tests are done | Research tests: |
| Поорна | study | | as part of the research on treatment for your condition. | Taking extra tubes of blood when you have regular blood tests (amount = 3 |
| | | | A measure of nutritional status will be obtained via a hand grip measurement with the JAMAR dynamometer. | tablespoons). Collecting urine in a container. Collecting stool in a container. |
| | | | Blood and urine for testing to see why alcohol caused your body to react in this way. These tests are done as part of the standard treatment for your condition. | |

The inflammation and liver markers in this study are designed for research, not for medical purposes. They are not useful for finding problems or diseases. Even though the researchers are not looking at your inflammation and liver markers to find or treat a medical problem, you will be told if they notice something unusual. You and your regular doctor can decide together whether to follow up with more tests or treatment. Because the inflammation and liver markers done in this study are not for medical purposes, the research results will not be sent to you or to your regular doctor. Your anonymous sample will be sent to coordinating research centers outside of UT Southwestern who are studying your disease. Your sample will be made anonymous by removing any identifiable information about you before it is shared with investigators outside of UT Southwestern.

#### Study Procedures by Study Day:

The procedures and evaluations are outlined below.

#### Screenina:

Complete screening will occur once the informed consent has been obtained as described above. Individuals who are not eligible for the study will be given the option for the same follow-up without the study medicine.

The study subject's general health and study information include:

- Signed consent
- Other routine information including sex, date of birth, race and ethnic group (Hispanic or not).
- Medicine history over the past 30 days, including prescribed and over-the-counter ones, herbal remedies, vitamins and minerals.
- Alcohol in the past 60 days and for the years before.

CONTINUE SELECT OF THE PROPERTY OF THE PROPERT

- Drawing blood for blood counts, clotting, and chemistry tests for the liver, pancreas and kidneys; female study subjects will have a pregnancy test. These are standard tests for your condition. The total amount of blood for these tests is about 7 tablespoons.
- Physical examination, including height, weight, and vital signs (blood pressure, pulse, breathing and temperature)
- Imaging of the abdomen.

#### Assessments:

#### Study day 0

- Record health history and review alcohol use.
- Standard of care laboratory studies (chemistry, blood count, clotting, urine, infection including tuberculosis testing)
- Tests for fluid in belly, if it is there
- Urine, blood (3 tablespoons) and stool testing for research.
- Nutritional Assessment with a hand grip measurement.
- Make a list of all medicines including those purchased over the counter, from health food stores and other remedies.
- Check blood pressure, pulse, temperature and breathing (vital signs) and physical exam.

## Procedures for storing of extra or left over samples

Samples of your blood and urine will be frozen and stored so that the researchers can test for any new inflammation or liver markers that are developed.

- Samples will be labeled with a study number, not with your name or other personal number.
- The key for study numbers will be kept in your medical record in a special section for research study information.
- The anonymous samples will be sent to Cleveland Clinic for storage
- The Principal Investigators will decide where and how the remaining samples will be processed
- Samples may be sent to other scientists for studies approved by their local IRB's to further understand this disease.

## What are the risks of the study?

#### **Psychological Stress**

Some of the questions we will ask you about your personal habits, as part of this study, may make you feel uncomfortable. You may refuse to answer any of the questions, take a break or stop your participation in this study at any time.

#### Loss of Confidentiality

Any time information is collected; there is a potential risk for loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

## Risks of Blood Drawing

Risks associated with drawing blood from your arm include minimal discomfort and/or bruising. Infection, excess bleeding, clotting, and/or fainting also are possible, although unlikely. You will have You will have 6 tablespoons of blood collected because you are in this research study, in

DO NOT DISCLOSE




addition to the tests that you need to take care of your health (another 13 tbspns over the 6 months).

## How will risks be minimized or prevented?

Potential risks and discomforts will be minimized to the greatest extent possible by appropriate training of all researchers and study personnel, monitoring you closely, withdrawal from the study upon evidence of difficulty or an adverse event; referral for treatment, counseling or other necessary follow-up.

#### What will my responsibilities be during the study?

While you are part of this study, the researchers will follow you closely to determine whether there are problems that need medical care. It is your responsibility to do the following:

- · Ask questions about anything you do not understand.
- Follow the researchers' instructions.
- Let the researchers know if your telephone number or address changes.

## If I agree to take part in this research study, will I be told of any new risks that may be found during the course of the study?

Yes. You will be told if any new information becomes available during the study that could cause you to change your mind about continuing to participate or that is important to your health or safety.

#### What should I do if I think I am having problems?

If you have unusual symptoms, pain, or any other problems while you are in the study, you should report them to the researchers right away. Telephone numbers where they can be reached are listed on the first page of this consent form. If you have a sudden, serious problem, like difficulty breathing or severe pain, go to the nearest hospital emergency room, or call 911 (or the correct emergency telephone number in your area). Tell emergency personnel about any medications you are taking, including any medications you are taking for this study.

#### What are the possible benefits of this study?

If you agree to take part in this study, the researchers cannot guarantee that you will benefit from participation in this research.

We hope the information learned from this study will benefit others with inflammation of the liver from alcohol. Information gained from this research could lead to treatment with lower risks of dying in the first 6 months after being admitted to the hospital for hepatitis from alcohol.

#### What options are available if I decide not to take part in this research study?

You do not have to participate in this research to receive care for your medical problem.

#### Will I be paid if I take part in this research study?

There are no funds available to pay for parking expenses, transportation to and from the research center, lost time away from work etc., lost wages, or child care expenses.

Will my insurance provider or I be charged for the costs of any part of this research study? No. Neither you, nor your insurance provider, will be charged for anything done only for this research study. However, the standard medical care for your condition (care you would have received whether or not you were in this study) is your responsibility (or the responsibility of your

DO NOT DISCLOSE

Study ID: STU 092012-012 Date Approved: 9/13/2017




insurance provider or governmental program). You will be charged, in the standard manner, for any procedures performed for your standard medical care.

## What will happen if I am harmed as a result of taking part in this study?

It is important that you report any illness or injury to the research team listed at the top of this form immediately. Compensation for an injury resulting from your participation in this research is not available from the University of Texas Southwestern Medical Center or Parkland Health & Hospital System. You retain your legal rights during your participation in this research

## Can I stop taking part in this research study?

Yes. If you decide to participate and later change your mind, you are free to stop taking part in the research study at any time. If you decide to stop taking part in this research study, it will not affect your relationship with the UT Southwestern staff or doctors. Whether you participate or not will have no effect on your legal rights or the quality of your health care.

## If I agree to take part in this research study, can I be removed from the study without my consent?

Yes. The researchers may decide to take you off this study if:

- The researchers believe that participation in the research is no longer safe for you.
- You are unable to follow the researcher's instructions.

## Will my information be kept confidential?

Medical information collected during this study and the results of any test or procedure done may be included in your medical record and this information may be available to health care providers and authorized persons including your insurance company.

You should know that certain organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- Cleveland Clinic, University of Louisville, University of Massachusetts, NIH
- Representatives of government agencies, like the U.S. Food and Drug Administration (FDA), involved in keeping research safe for people; and
- The UT Southwestern Institutional Review Board.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by the U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

In addition to this consent form, you will be asked to sign an "Authorization for Use and Disclosure of Protected Health Information." This authorization will give more details about how your information will be used for this research study, and who may see and/or get copies of your information.

## Are there procedures I should follow after stopping participation in this research?

Yes. If you, the researchers, or the sponsor stops your participation in the research, you may be asked to do the following:

- Let the researchers know immediately that you wish to withdraw from the research.
- Return to the research center for tests that may be needed for your safety.

DO NOT DISCLOSE




• Discuss your future medical care, if any, with the researchers and/or your personal doctor.

## Whom do I call if I have questions or problems?

For questions about the study, contact Dr. Mitchell at 214-648-4570 during regular business hours and at 214-648-3111 after hours and on weekends and holidays.

For questions about your rights as a research participant, contact the UT Southwestern Institutional Review Board (IRB) Office at 214-648-3060.

THE CONTROL OF THE CO

 DO NOT DISCLOSE

#### **SIGNATURES:**

#### YOU WILL BE GIVEN A COPY OF THIS CONSENT FORM TO KEEP.

Your signature below certifies the following:

- You have read (or been read) the information provided above.
- You have received answers to all of your questions and have been told who to call if you
  have any more questions.
- You have freely decided to participate in this research.
- You understand that you are not giving up any of your legal rights.
- You understand that a copy of this signed consent document, information about this study
  and the results of any test or procedure done may be included in your medical record and
  this information may be available to health care providers and authorized persons
  including your insurance company.

| Participant's Name (printed) | |
|--------------------------------------------|-------------|
| Participant's Signature | Date & Time |
| Name of person obtaining consent (printed) | |
| Signature of person obtaining consent | Date & Time |

DO NOT BIOCH COF



## The University of Texas Southwestern Medical Center at Dallas Parkland Health & Hospital System

#### **CONSENT TO PARTICIPATE IN RESEARCH**

Title of Research: Novel therapies in moderately severe alcoholic hepatitis

Funding Agency/Sponsor: NIH (funded)

Study Doctors: Mack Mitchell, M.D.

Lisa Casey, M.D. Jennifer Cuthbert, M.D.

You may call these study doctors or research personnel during regular office hours at 214-648-4570. At other times, you may call them at 214-648-3111 and tell them that you need to contact your study doctors. Have the study information with you when you call after hours so that the hospital operators know who to contact.

#### Instructions:

Please read this consent form carefully and take your time making a decision about whether to participate. As the researchers discuss this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. The purpose of the study, risks, inconveniences, discomforts, and other important information about the study are listed below. If you decide to participate, you will be given a copy of this form to keep.

#### Why is this study being done?

This study is being done to follow what happens to the liver in response to inflammation from alcohol by collecting and testing research samples. The research studies will not improve the health of your liver.

## Why is this considered research?

This is a research study because the tests are not routine for patients with liver problems.

## The following definitions may help you understand this study:

- Standard medical care means the regular care you would receive from your personal doctor if you choose not to participate in this research.
- Researcher means the study doctors and research personnel at the University of Texas Southwestern Medical Center at Dallas and its affiliated hospitals.

#### Why am I being asked to take part in this research study?

You are being asked to take part in this study because you have an inflamed liver (hepatitis) that your doctors' think is from your body's reaction to alcohol.

#### Do I have to take part in this research study?"

No. You have the right to choose whether you want to take part in this research study. If you decide to participate and later change your mind, you are free to stop participation at any time. If you decide not to take part in this research study it will not change your legal rights or the quality of health care that you receive at this center.

### How many people will take part in this study?

About 50 people will take part in the medication study at UT Southwestern or Parkland Health and Hospital System. This study also is taking place at a number of other medical facilities around the country. There will be



a total of 130 people participating in this research study throughout the United States. People who don't want to take a medication can be part of the research by participating in the new tests.

#### What is involved in the study?

If you volunteer to take part in this research study, you will be asked to sign this consent form and will have the following tests and procedures. Some of the procedures may be part of your standard medical care, but others are being done solely for the purpose of this study.

## Screening Procedures

To help decide if you qualify to be in this study, the researchers will ask you questions about your health, including medications you take, your diet and habits. They will also get information from your medical record.

#### Procedures and Evaluations during the Research

All study subjects will receive the standard medical care used for patients with hepatitis from your body's reaction to alcohol. This includes:

- 1. A good diet while in the hospital and recommendations for what to eat at home
  - a. Lots of fresh vegetables, fruits, chicken, fish
  - b. Vitamins and other special nutrition if needed
- 2. Help with avoiding alcohol in the future
  - a. Counselors
  - b. Psychologists
  - c. Rehabilitation assistance
- 3. Only take medications prescribed by your doctors. Do not take any medication or diet supplement or over-the-counter remedy without checking with a study doctor or nurse. Avoid all pain medicines that have high risk associated with them because of liver disease.
  - a. Aspirin and over the counter medications like ibuprofen Motrin®, Aleve® can damage the kidneys with as little as one tablet
  - b. Stronger pain medicines that contain codeine or a similar agent can cause confusion related to liver disease
  - c. Acetaminophen (Tylenol®) can directly cause liver damage
- 4. Treatment for any complications that can occur
  - a. Antibiotics for infections
  - b. Treatment for diarrhea or constipation or nausea and vomiting if they occur
- 5. Blood drawing to follow the changes in your liver.
- 6. Follow-up in the regular outpatient liver clinic, after you leave the hospital, until your liver has completely recovered. The number of visits depends on how quickly you get better. This is likely to be:
  - a. 1 week after leaving the hospital
  - b. 1-2 visits in the next month
  - c. 1-2 visits in the next 2-4 months, depending on how quickly you get well
  - d. A final clinic visit after 6 months



In addition, the following special, extra studies will be done for research purposes when you come into clinic:

| Where | When | What | How |
|---|---|---|---|
| In<br>hospital | First day of the study | Inflammation markers and liver markers will be measured. These tests are done as part | Research tests: |
| rioopitai | tile stady | of the research on treatment for your condition. | Taking extra tubes of blood when you have regular blood tests (amount = 3 |
| | | Blood and urine for testing to see why alcohol caused your body to react in this way. These tests are done as part of the standard treatment for your condition. | tablespoons). Collecting urine and stool in a container. |
| In<br>hospital<br>or in | Day 7 | Inflammation markers and liver markers will<br>be measured. These tests are done as part<br>of the research on treatment for your | Research tests: Taking extra tubes of blood |
| clinic | | condition. | when you have regular blood<br>tests (amount = 2 |
| | | Blood and urine for testing to see why alcohol caused your body to react in this way. These tests are done as part of the standard treatment for your condition. | tablespoons). Collecting urine in a container. |
| In clinic | 1 month<br>3 months | Inflammation markers and liver markers will be measured. These tests are done as part | Research tests: |
| | 6 months | of the research on treatment for your condition. | Taking extra tubes of blood when you have regular blood tests (amount = 3 |
| | | A blood test to see if your gut is leaky. This test is part of the research on treatment for your condition. | tablespoons). Collecting urine and stool in a container. |
| | | Blood and urine for testing to see why alcohol caused your body to react in this way. These tests are done as part of the standard treatment for your condition. | |

The inflammation and liver markers in this study are designed for research, not for medical purposes. They are not useful for finding problems or diseases. Even though the researchers are not looking at your inflammation and liver markers to find or treat a medical problem, you will be told if they notice something unusual. You and your regular doctor can decide together whether to follow up with more tests or treatment. Because the inflammation and liver markers done in this study are not for medical purposes, the research results will not be sent to you or to your regular doctor. Your anonymous sample will be sent to coordinating research centers outside of UT Southwestern who are studying your disease. Your sample will be made anonymous by removing any identifiable information about you before it is shared with investigators outside of UT Southwestern.

## Study Procedures by Study Day:

A summary of evaluations is located in the schedule of events table provided at the end of this section. The procedures and evaluations are outlined below.

#### Screening:

Complete screening will occur once the informed consent has been obtained as described above. Individuals who are not eligible for the study will be given the option for the same follow-up without the study medicine.



The study subject's general health and study information include:

- Signed consent
- Other routine information including sex, date of birth, race and ethnic group (Hispanic or not).
- Medicine history over the past 30 days, including prescribed and over-the-counter ones, herbal remedies, vitamins and minerals.
- Alcohol in the past 60 days and for the years before.
- Drawing blood for blood counts, clotting, and chemistry tests for the liver, pancreas and kidneys; female study subjects will have a pregnancy test. These are standard tests for your condition. The total amount of blood for these tests is about 7 tablespoons.
- Physical examination, including height, weight, and vital signs (blood pressure, pulse, breathing and temperature)
- Imaging of the abdomen.

## Assessments at baseline and during study:

Study Procedures by Study Day:

A summary is in the table at the end of this section.

Study day 0 – start (within 24 hours of study beginning)

- Record health history and review alcohol use.
- Standard of care laboratory studies (chemistry, blood count, clotting, urine, infection including tuberculosis testing)
- Tests for fluid in belly, if it is there
- Urine, blood (3 tablespoons) and stool testing for research.
- Make a list of all medicines including those purchased over the counter, from health food stores and other remedies.
- Nutritional Assessment with a hand grip measurement.
- Check blood pressure, pulse, temperature and breathing (vital signs) and physical exam.

#### Study day 1 – time zero

Standard blood tests for your condition (1 tablespoon)

### Study day 2:

- Inpatient assessment to include:
  - Review health history for changes.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine and ½ tablespoon of blood).
  - 24 hour urine collection.
- Standard blood tests for your condition (1½ tablespoons)

#### Study days 3-6:

- If study subject remains inpatient or has outpatient visit:
  - Review health history for changes. .
  - List all medicines
  - Check vital signs and physical exam
- Standard blood tests for your condition (1 tablespoon)

#### Study day 7:

- Inpatient assessment or outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines



- Check vital signs and physical exam
- Research studies (urine and 1 tablespoon of blood).
- Standard and research blood tests (2 tablespoons)
- Nutritional Assessment with a hand grip measurement.

#### Study days 8-14:

- If study subject remains inpatient or has outpatient visit:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
- Standard blood tests for your condition (1 tablespoon)

#### Study days 15-27:

- If study subject remains inpatient or has a clinically indicated outpatient visit:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
- Stop taking the injection once a day
- Standard blood tests for your condition (1 tablespoons)

## Study day 28:

- Inpatient assessment or outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine and ½ tablespoon blood).
- Standard and blood tests for your condition (1½ tablespoon)
- Nutritional Assessment with a hand grip measurement.

#### Study day 29 to 2 months:

- If study subject remains inpatient during this interval or completes clinically indicated outpatient visit during this time, the following data will be recorded:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Standard blood tests for your condition (1 tablespoons)

#### Study 3 months ± 2 weeks:

- Inpatient assessment or outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine, stool and ½ tablespoon blood).
- Standard blood tests for your condition (1½ tablespoon)

## Study 4, 5 months ± 2 weeks:

- If study subject remains inpatient or completes clinically indicated outpatient visit during this time, the following will be done:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam



• Standard blood tests for your condition (1 tablespoons)

#### Study 6 months ± 2 weeks:

- Complete abdominal ultrasound.
- Inpatient assessment or outpatient clinic visit to include:
  - Review health history for changes. Review alcohol intake.
  - List all medicines
  - Check vital signs and physical exam
  - Research studies (urine, ½ tablespoon blood and stool).
- Standard blood tests for your condition (1½ tablespoons)
- Nutritional Assessment with a hand grip measurement.

#### Procedures for storing of extra or left over samples

Samples of your blood and urine will be frozen and stored so that the researchers can test for any new inflammation or liver markers that are developed.

- Samples will be labeled with a study number, not with your name or other personal number.
- The key for study numbers will be kept in your medical record in a special section for research study information.
- The anonymous samples will be sent to Cleveland Clinic for storage
- The Principal Investigators will decide where and how the remaining samples will be processed
- Samples may be sent to other scientists for studies approved by their local IRB's to further understand this disease.

#### How long can I expect to be in this study?

The study is for a total of 6 months, first as an inpatient and then as an outpatient for a total of 6 months. You can choose to stop participating for any reason at any time. However, if you decide to stop participating in the study, we encourage you to tell the researchers. You will be asked if you are willing to complete some study termination tests.



Page 6 of 11

| Purpose | Test | Day 0 | Day 2 – 6* | Day 7 | Day<br>8 – 27* | Day 28 | 2 mos* | 3 mos | 4 mos* | 5 mos* | 6 mos |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Standard | General health and liver questions | х | х | х | х | х | х | Х | х | х | Х |
| | Questions about drinking alcohol | х | х | х | х | х | х | х | х | х | х |
| | Physical exam | х | х | х | х | х | х | х | х | х | х |
| Blood | Liver tests | х | х | х | х | х | х | х | х | х | х |
| | Tests of chemicals and kidneys | х | х | х | х | х | х | Х | х | х | х |
| | Blood count | х | х | х | х | х | х | х | х | х | х |
| | Cholesterol test | х | | | | | | | | | х |
| | Pancreas tests | x | | | | | | | | | |
| | Tests for viruses and bacteria | x | | | | | | | | | |
| | TB skin test | x | | | | | | | | | |
| Urine | Urine tests | х | | | | | | | | | |
| | Poisons | х | | | | | | | | | |
| Fluid | Belly fluid chemicals and infection | x | | | | | | | | | |
| Stool | Infection tests | х | | | | | | | | | |
| Imaging | Ultrasound of belly | x | | | | | | | | | х |
| Research | Gut leakiness | x | | | | х | | х | | | х |
| | Zinc levels | x | | | | х | | х | | | х |
| | Stool bacteria tests | х | | | | | | х | | | х |
| | Inflammation tests | х | x-day 2 | х | | х | | х | | | x |

<sup>\*</sup> if clinically indicated



## What are the risks of the study?

## Psychological Stress

Some of the questions we will ask you about your personal habits, as part of this study, may make you feel uncomfortable. You may refuse to answer any of the questions, take a break or stop your participation in this study at any time.

#### Loss of Confidentiality

Any time information is collected; there is a potential risk for loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

## Risks of Blood Drawing

Risks associated with drawing blood from your arm include minimal discomfort and/or bruising. Infection, excess bleeding, clotting, and/or fainting also are possible, although unlikely. You will have 6 tablespoons of blood collected because you are in this research study, in addition to the tests that you need to take care of your health (another 13 tbspns over the 6 months).

#### How will risks be minimized or prevented?

Potential risks and discomforts will be minimized to the greatest extent possible by appropriate training of all researchers and study personnel, monitoring you closely, withdrawal from the study upon evidence of difficulty or an adverse event; referral for treatment, counseling or other necessary follow-up.

#### What will my responsibilities be during the study?

While you are part of this study, the researchers will follow you closely to determine whether there are problems that need medical care. It is your responsibility to do the following:

- Ask guestions about anything you do not understand.
- Keep your appointments.
- Follow the researchers' instructions.
- Let the researchers know if your telephone number or address changes.
- Tell the researchers before you take any new medication, even if it is prescribed by another doctor for a different medical problem or something purchased over the counter.
- Tell your regular doctor about your participation in this study.
- Carry information about contacting the study doctors in your purse or wallet.
- Report to the researchers any injury or illnesses while you are on study, even if you do not think they are related.

## If I agree to take part in this research study, will I be told of any new risks that may be found during the course of the study?

Yes. You will be told if any new information becomes available during the study that could cause you to change your mind about continuing to participate or that is important to your health or safety.



## What should I do if I think I am having problems?

If you have unusual symptoms, pain, or any other problems while you are in the study, you should report them to the researchers right away. Telephone numbers where they can be reached are listed on the first page of this consent form. If you have a sudden, serious problem, like difficulty breathing or severe pain, go to the nearest hospital emergency room, or call 911 (or the correct emergency telephone number in your area). Tell emergency personnel about any medications you are taking.

#### What are the possible benefits of this study?

If you agree to take part in this study, there may be direct benefits to you. The researchers cannot guarantee that you will benefit from participation in this research.

We hope the information learned from this study will benefit others with inflammation of the liver from alcohol. Information gained from this research could lead to treatment with lower risks of dying in the first 6 months after being admitted to the hospital for hepatitis from alcohol.

#### What options are available if I decide not to take part in this research study?

You do not have to participate in this research to receive care for your medical problem. Instead of being in this study, you have the following option:

Being treated with standard medical care

Please talk to the researchers or your personal doctor about these options.

#### Will I be paid if I take part in this research study?

There are no funds available to pay for parking expenses, transportation to and from the research center, lost time away from work etc., lost wages, or child care expenses.

Will my insurance provider or I be charged for the costs of any part of this research study? No. Neither you, nor your insurance provider, will be charged for anything done only for this research study. However, the standard medical care for your condition (care you would have received whether or not you were in this study) is your responsibility (or the responsibility of your insurance provider or governmental program). You will be charged, in the standard manner, for any procedures performed for your standard medical care.

#### What will happen if I am harmed as a result of taking part in this study?

It is important that you report any illness or injury to the research team listed at the top of this form immediately. Compensation for an injury resulting from your participation in this research is not available from the University of Texas Southwestern Medical Center or Parkland Health & Hospital System. You retain your legal rights during your participation in this research

## Can I stop taking part in this research study?

Yes. If you decide to participate and later change your mind, you are free to stop taking part in the research study at any time. If you decide to stop taking part in this research study, it will not affect your relationship with the UT Southwestern staff or doctors. Whether you participate or not will have no effect on your legal rights or the quality of your health care.



## If I agree to take part in this research study, can I be removed from the study without my consent?

Yes. The researchers may decide to take you off this study if:

- The researchers believe that participation in the research is no longer safe for you.
- You are unable to follow the researcher's instructions.

## Will my information be kept confidential?

Medical information collected during this study and the results of any test or procedure done may be included in your medical record and this information may be available to health care providers and authorized persons including your insurance company.

You should know that certain organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- · Cleveland Clinic, University of Louisville, University of Massachusetts, NIH
- Representatives of government agencies, like the U.S. Food and Drug Administration (FDA), involved in keeping research safe for people; and
- The UT Southwestern Institutional Review Board.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by the U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

In addition to this consent form, you will be asked to sign an "Authorization for Use and Disclosure of Protected Health Information." This authorization will give more details about how your information will be used for this research study, and who may see and/or get copies of your information.

#### Are there procedures I should follow after stopping participation in this research?

Yes. If you, the researchers, or the sponsor stops your participation in the research, you may be asked to do the following:

- Let the researchers know immediately that you wish to withdraw from the research.
- Return to the research center for tests that may be needed for your safety.
- Discuss your future medical care, if any, with the researchers and/or your personal doctor.



## Whom do I call if I have questions or problems?

For questions about the study, contact Dr. Mitchell at 214-648-4570 during regular business hours and at 214-648-3111 after hours and on weekends and holidays.

For questions about your rights as a research participant, contact the UT Southwestern Institutional Review Board (IRB) Office at 214-648-3060.

#### **SIGNATURES:**

#### YOU WILL BE GIVEN A COPY OF THIS CONSENT FORM TO KEEP.

Your signature below certifies the following:

- You have read (or been read) the information provided above.
- You have received answers to all of your questions and have been told who to call if you have any more questions.
- You have freely decided to participate in this research.
- You understand that you are not giving up any of your legal rights.
- You understand that a copy of this signed consent document, information about this study
  and the results of any test or procedure done may be included in your medical record and
  this information may be available to health care providers and authorized persons
  including your insurance company.

| Participant's Name (printed) | |
|--------------------------------------------|-------------|
| Participant's Signature | Date & Time |
| Name of person obtaining consent (printed) | |
| Signature of person obtaining consent | Date & Time |

Page 11 of 11

